CLINICAL TRIAL: NCT05506657
Title: Early Intervention to Promote Return to Work for People With Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-1171-21A
Record Dates: First submitted 2022-01-19; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: employment; vocational rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- State Counselor-Coordinated Services (Other): In this program, services are coordinated by a counselor employed by the New Jersey State Division of Vocational Rehabilitation Services (NJDVRS), a state-based agency that assists people with disabilities who are interested in pursuing employment. While the participant is in inpatient rehabilitation or soon after their discharge, a member of the research team will assist them in completing the necessary documentation to apply for services from this agency. Services for which they are eligible will be provided directly through NJDVRS.
  Interventions: Other: State Counselor-Coordinated Services
- Center Facilitator-Coordinated Services (Other): In this program, services are coordinated by a facilitator who is employed by Kessler Institute for Rehabilitation and works cooperatively with NJDVRS. The facilitator will begin working with the participant during inpatient rehabilitation, or soon after discharge, depending on when they enroll in the study. Some services for which they are eligible will be provided through NJDVRS and others will be provided to them by the facilitator.
  Interventions: Other: Center Facilitator-Coordinated Services

INTERVENTIONS:
Other: State Counselor-Coordinated Services — A counselor affiliated with the New Jersey State Division of Vocational Rehabilitation Services coordinates services that consider the participant's condition, needs and goals. Services participants may receive include:
  * Education on programs designed to help people with spinal cord injury or brain injury pursue employment.
  * Advice and guidance from professional counselors who have special training in helping people with disabilities pursue employment.
  * Help completing applications for services.
  * Assistance communicating with my employer about my needs and ways to accommodate them.
  * Referrals to and services from other health care or technology providers.
  Arms: State Counselor-Coordinated Services
Other: Center Facilitator-Coordinated Services — A facilitator affiliated with Kessler Institute for Rehabilitation coordinates services that consider the participant's condition, needs and goals. Services participants may receive include:
  * Education on programs designed to help people with spinal cord injury or brain injury pursue employment.
  * Advice and guidance from professional counselors who have special training in helping people with disabilities pursue employment.
  * Help completing applications for services.
  * Assistance communicating with my employer about my needs and ways to accommodate them.
  * Referrals to and services from other health care or technology providers.
  Arms: Center Facilitator-Coordinated Services

SUMMARY:
For many people with spinal cord injury, seeking employment after injury is an important goal. There are services available to help people with disabilities. However, the best ways to coordinate and deliver these services are not yet known. This project will compare two ways of coordinating and delivering services that are designed to help people with spinal cord injury obtain employment.

DETAILED DESCRIPTION:
Employment is important for financial security, social connection, and life satisfaction. Unfortunately, rates of unemployment remain high among people with spinal cord injury (SCI). To help address this challenge, the Northern New Jersey Spinal Cord Injury System (NNJSCIS) is conducting a single-site, randomized, controlled trial to compare two programs intended to increase rates of employment among people with SCI. The project will enroll 162 recently injured adults with SCI who are interested in becoming employed or returning to work and will compare different ways of delivering employment-related services in the first year after injury. Services will begin in inpatient rehabilitation and may include education, therapy, equipment provision, counseling, and other interventions. Information about employment status, earnings, community participation, and health will be collected through a combination of questionnaires and databases. Participants and service providers will also share their impressions of the programs via survey and focus groups. Analyses will examine the rate of participants employed at 1 year in each group, time to employment, earnings, community participation, and other aspects of well-being. Findings from this study will be used to determine which ways of delivering services are most effective in enabling employment by 1 year after injury, and to provide information to help other rehabilitation centers adopt effective programs.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 to 62
* a neurological impairment secondary to an SCI that occurred less than 12 months prior to enrollment
* receiving inpatient rehabilitation at Kessler Institute for Rehabilitation (KIR)
* community living in the state of NJ after discharge from KIR
* have a goal to pursue competitive integrated employment or education/retraining leading to competitive integrated employment

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Employment Status (Percent Employed) | 12-months post-enrollment
  Proportion of participants in each group in competitive employment.

SECONDARY OUTCOMES:
Employment Efficiency (Median Time to Employment) | 12-months post-enrollment
  Median number of months from date of enrollment to date of competitive integrated employment; obtained through self-report.
Income | 12-months post-enrollment
  Earnings within the first 12 months post-enrollment as obtained from New Jersey Unemployment Insurance (UI) data.
Satisfaction with Life Scale (SWLS) | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  5 item (2 minute) scale that provides global measure of life satisfaction.
International SCI Quality of Life Basic Data Set | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  3 item (~1 minute) assessment of satisfaction with life as a whole, physical health, psychological health.
Craig Handicap Assessment and Reporting Technique (CHART) | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  Subscales examine several objective physical independence, cognitive independence, mobility, occupation, social integration, and economic self-sufficiency; includes personal care assistance use.
Spinal Cord Injury Quality of Life: Satisfaction with Social Roles and Activities (SCI-QoL) | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  10 item short form (<5 minutes) examining extent of satisfaction or disappointment with social roles and activities; complements CHART.
Patient Health Questionnaire (PHQ-9) | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  Measure of depressive symptomology (9 items; 3 minutes).
Spinal Cord Injury Quality of Life: Self-Esteem | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  8 item (<5 minute) short form; assesses emotional, evaluative, and cognitive perceptions of personal competence and worth.
Spinal Cord Injury Quality of Life: Independence | Assessed at 1 month (baseline), 6, and 12 months post-enrollment.
  8 item (<5 minute) short form.
Exit Survey | 12-months post-enrollment
  Includes rating scale and open-ended items pertaining to satisfaction with the program and suggestions for optimization of the programs.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Dyson-Hudson, M.D., Principal Investigator — Kessler Foundation; John O'Neill, Ph.D., Principal Investigator — Kessler Foundation

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD), except if/when limited by data use agreements established with the New Jersey Department of Labor, will be shared via the Interuniversity Consortium for Political and Social Research (ICPSR), the preferred data repository for the National Institute on Disability, Independent Living, and Rehabilitation Research. Data shared via ICPSR will include data from measures collected at baseline and follow-ups for purposes of sample characterization and/or outcomes assessment. All data will be de-identified and labeled with subject identification numbers established for the study rather than names or initials.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made available within 6-12 months of the completion of the study and will remain available indefinitely.
Access Criteria: Requests for data access will be coordinated through the Interuniversity Consortium for Political and Social Research (ICPSR) according to their established procedures.
URL: https://www.icpsr.umich.edu/web/pages/